CLINICAL TRIAL: NCT02589574
Title: Improving Influenza Vaccination Rates in Nurses Through Electronic Text Message Reminders : a Randomised Controlled Trial
Brief Title: Improving Influenza Vaccination Rates in Nurses Through Text Message Reminders : a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Angela Y.Y. Cheung, Doctorate degree student, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW15-383
Record Dates: First submitted 2015-10-15; First posted 2015-10-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Subjects of the control group will receive the usual announcement on the dates and times of offering free influenza vaccination, and reminder from hospital, and access to informational flyers posted at the hospital
- Intervention (Experimental): Subjects of the intervention group besides the usual information same as those stated in the control group, will receive four reminders on dates and details for free influenza vaccine. Together with the reminder, electronic text messages of educational information will be received
  Interventions: Other: electronic text message

INTERVENTIONS:
Other: electronic text message — Besides the reminder of the free vaccination, the messages included information that vaccination reduces the personal risk of influenza illness. It also reduces the risk to infect patients and family members. It is also the social expectation on and professional as well as personal responsibility of nurses in protecting own selves and their patients from contacting influenza.
  it is a safe vaccine. The reminders are developed with reference to promotion messages from Hospital Authority.
  Arms: Intervention

SUMMARY:
Influenza is an important cause of medical visits and worker absenteeism among healthy adults. Studies of healthcare providers vaccination programmes have reported a positive effect in lowering rates of influenza like illness and influenza related complication, hospitalisation and death. Nurses should receive influenza vaccination so that those patients who may come in contact with will not be infected by their nurses. However, the immunization rate among nurses is constantly low. Therefore, it is important to develop an intervention programmes to increase immunization of nurses. In some research on electronic text messaging in promoting public health showed potential of this communication system in preventive health behavioural change. With the use of this widely acceptable, accessible and convenient approach of communication, reminders of receiving influenza vaccination are sent to nurses involved in this study. At the same time, educational messages are sent to modify their perception on the positive effect of influenza vaccination, and therefore, motivate the nurses to receive the vaccination. The study will be conducted as a two-arm randomised controlled trial which the control and intervention groups will run concurrently. Nurses of a local hospital are invited to participate in this study. They will receive the usual announcement on the information of free influenza vaccination of the hospital. The participants of the intervention group will also receive text message reminders on details for free influenza vaccine and educational information. All communication occurred through secure, asynchronous electronic text messages. The reminders and educational information are developed with reference to promotion messages from the Department of Health under the framework of Health Belief Model so as to promote positive perception on influenza vaccination by the participants. Participants are invited to complete the pre and post questionnaires before and after the study period. The influenza vaccination status of the participants and their perception on influenza vaccination will be obtained. It is hypothesised that the participants receiving the reminders and educational information will more likely to receive influenza vaccine and perceived the influenza vaccination as important measure in protecting them from influenza. The participants of the intervention group will also receptive to electronic text messaging communication and education.

DETAILED DESCRIPTION:
The Study aims to evaluate the efficacy of text messaging reminders in promoting influenza vaccination among nurses in a Hong Kong local hospital. The primary outcome is the receipt of influenza vaccine by end of February 2016 as reported by the participants. The secondary outcomes include the proportion of participants seeking out influenza vaccination and the proportion of participants of intervention group receptive to electronic text messaging communication and education. According to a study by WHO in 2005, influenza vaccines offer approximately 70-90% protection against clinical diseases in healthy adults. Despite the recommendation suggested by the CHP of Hong Kong that vaccination should be received by the high risks groups such as healthcare providers including nurses, vaccination rate of nurses is remained low with the Annual Seasonal Influenza Uptake Rate at 14.41% in 2013 in Hong Kong. This finding corresponded to those overseas studies that the influenza vaccine rate of nurses was among the lowest of all healthcare providers.

Although numerous interventions have been employed to promote Influenza vaccination, the cost of these approaches are high whilst have not resulted in the large or long-lasting increase that has been desired. Moreover, there are factors that inhibit nurses from receiving vaccination. Studies showed that nurses perceived themselves low risk from influenza. Other reasons such as misunderstanding and myths about influenza can be acquired from the vaccine, concerns about the efficacy and side effects of vaccine, and lack of time or forgot.

Nurses also perceived there is absence of an immediate threat to their health, especially for the younger nurses. Hence, tend not to seek out influenza vaccination. A study found that one of the stipulated reasons nurses for choosing to be vaccinated against influenza was their concern about spreading the disease to their patients if the nurses got influenza, which was the second highest reason other than concern about getting influenza themselves. The findings coherence with the caring nature of persons who entered nursing. Other findings also found that recall system and educational information with the emphasis on recommended vaccination are ranked as the second and third most effective strategies to improve or maintain vaccination coverage.

Nowadays, using electronic reminder system is not new to nurses in Hong Kong. The implementation of Clinical Dash Board was introduced about 10 years ago and has been used to generate messages to alert nurses to deal with their varied unfinished clinical works as well as appointment of the patients under their care. At the same time, mobile technologies were considered by many to be the next frontier in health behaviour change because they were considered to be the vehicles to deliver personal and adaptive health information anywhere in real time. It is suggested by some researchers that electronic text messaging might hold a more promising result in serving as a reminder. There is a growing body of researches on text messaging for a range of health and mental health problems. However, none of these studies reported on receiving text messages in promoting vaccination uptake of nurses, the single largest group of healthcare providers who close encounter with people that are highly susceptible to influenza and other upper respiratory diseases. It is the intention of this study to look into the issue so as to evaluate the efficacy of text messaging reminders in promoting influenza vaccination among nurses.

Subjects of the study included qualified nurses who are employed in a Hong Kong local hospital, owned smart phones with electronic text messaging function, and are willing to provide their active mobile telephone numbers. However, qualified nurses who have already received influenza vaccination prior the commencement of vaccination period of 2015-16, or who have history of allergies to egg, chicken proteins or neomycin or any component of vaccine, or who have history of moderate to severe reaction to influenza vaccination, or who have history of Guillain-Barré Syndrome will be excluded.

As there is no randomised control trial study has been found from the literature that evaluate the effect of text messaging on increase influenza vaccine uptake of nurses, similar study with subject other than nurses was referred. With reference to other similar study, the overall vaccination rate among participants of both control and intervention groups ranged from 18.1% to 36.4% with the effect size of around 18%. Taking reference to the influenza vaccination uptake rate of the local hospital which this study is intended to be carried out was only 11.56% in the seasonal influenza period 2013-14, it is estimated that the vaccination rate of nurses in the intervention group of the proposed study would be 17%. Given α = 0.05, desired power = 0.8, by comparing two proportions, the number of subject in each group should be at least 247. Allowing a drop-out rate of 25%, 329 subjects in each group should be provided the desired power. Hence, a sample size with minimum of 658 shall be recruited into this study.

Upon received the approval from the Research Ethics Committee of the Hospital, email will be sent to the nurse managers of each department and ward of the local hospital to introduce the study. Appointment will be made with the individual nurse manager regarding the appropriate time to brief the nurses. It is planned to carry out the briefing session during the recommended period where most of the nurses will be available to attend. The investigator will provide verbal explanation and distribute the information sheets to the participants prior to the commencement of data collection. Participants are encouraged to clarify any queries related to the study. Participation in the study will be entirely voluntary and each participant has the right to withdraw or refuse to give information at any time during the study without incurring any penalties or deprivation of services. The purpose and procedure of the study as well as the risks and benefits of participation will be explained. With this understanding, the participants are invited to sign the written consent form. Attached with it, a self-administered questionnaire will be given to the participants to complete. The completed questionnaire can be returned to the investigator at the time of briefing. For those who completed the post-intervention questionnaire by telephone interview, a message will be texted to each of these subjects which can be used for redemption of a $10 cash coupon from the investigator.

This study will be conducted with the respect for the individual participant in accordance with the requirement of this study protocol and also the International Conference on Harmonisation E6 Good Clinical Practice and all applicable laws and regulations, including without limitation, data privacy laws, clinical trial disclosure laws, and regulations.

Subjects will be recruited from November 2015 followed by data collection via pre and post questionnaires survey by March 2016. A randomizer, who will not be involved in any part of the study, will develop a randomised intervention allocation sequence using random block sizes of two, four, and six. Sequentially numbered, opaque and sealed envelopes containing assignment information will then be prepared and kept by the investigator who will responsible for participant recruitment. When informed written consent is obtained, the investigator will select the next envelope in the sequence to decide the intervention allocation.

During the study period, four electronic text messages will be sent to intervention group participants. Messages contain educational information such as the fact that during epidemic, nurses who are in close contact with high risk patients, are more likely to get an influenza infection; vaccination reduces the personal risk of influenza illness and also reduces the risk to infect patients and family members; by reducing the chance of sick leave due to influenza-like illnesses, vaccination can in turn reduce work pressure; lastly it is also the social expectation on the professional as well as personal responsibility of nurses in protecting own selves and their patients from contacting influenza.

The text messages on reinforcing the fact that influenza is dangerous for the nurses and for the patients will also mention. Therefore, any potential side effect is no reason for not being vaccinated. Vaccination cannot cause influenza infection nor reduce immunity. Influenza vaccine is a safe vaccine.

The messages will be sent to the intervention group participants on a weekly basis for 4 weeks. All communication occurred through a secure, asynchronous electronic text messages apps. The education information is developed with reference to promotion messages from Department of Health under the framework of health belief model which four constructs on which individuals base their perceptions, namely perceived benefit, perceived barriers, perceived susceptibility, and perceived seriousness of illness or threat.

Data analysis will be started in April 2016 and by August 2016, report will be generated and findings will be disseminated. A research assistant, who will not be involved in participant recruitment and will be blinded to the participants' intervention allocation, is responsible for the assessment of the study outcomes. The influenza vaccination status of the participants will be obtained through telephone follow up by the research assistant.

The project will be evaluated by quantitative method. All participants will be asked to complete the questionnaires before and after the influenza season. The questionnaires will include the participants' vaccination status, their perception on influenza vaccination, their history of contacting influenza or experiencing influenza-like illnesses, and their experience and perceptions of the effectiveness of the use of electronic text message reminder in promoting health intervention. The study analyses will be conducted using SPSS 21.0. The significant level selected for all analyses was P ≤ 0.05. Descriptive baseline characteristics of the groups were tabulated as means and standard deviations or proportions. Differences in demographic characteristics between the intervention and control group will be analysed using t-test for continuous data and chi-square tests for categorical data. The primary concern of the study will compare the influenza vaccine uptake in the two study groups. For the primary outcome on influenza vaccine uptake, the investigators will calculate risk differences (RD) and relative risks (RR) with their corresponding 95% confidence intervals (95%CI). The efficacy analysis will be performed in accordance with the intention-to-treat principle that with missing data taken as no vaccination received. Differences in the facilitators will also be compared, again using chi-square test.

To protect the privacy of the participants, the data would be handled and stored by the investigator in a confidential way during and after the completion of the study. All the data set would be handled in line with Hospital's policy in handling, storage and destruction of confidential records. They would be kept by the investigator in a cabinet with lock which is located in her office. Electronic data would be saved in secured computer in the investigator's office with restricted access. Access to the data would only be made with the approval from the Principal Investigator, hence, confidentiality and anonymity will be assured.

ELIGIBILITY:
Inclusion Criteria:

1. qualified nurses who are employed in the local hospital during the period of study
2. owned smart phones with electronic text messaging function
3. willing to provide their active mobile telephone numbers
4. who have already received influenza vaccination prior to the commencement of the study period or those have history of allergy to flu vaccine will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The receipt of an influenza vaccine dose by Feb 2016 as reported by the participants | up to 5 months

SECONDARY OUTCOMES:
The proportion of participants seeking out influenza vaccination | up to 5 months
The proportion of participants of intervention group receptive to electronic text messaging communication and education | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Tarrant, PhD, Study Director — The University of Hong Kong
Locations (1):
- United Christian Hospital, Hong Kong, China